CLINICAL TRIAL: NCT05224076
Title: The Changing COVID-19 Landscape: A Feasibility Study to Capture Momentary Residential Environmental Exposures and Asthma Symptoms in Adults
Brief Title: Home Air Quality Impact for Adults With Asthma
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Other Study IDs: STUDY00145830; R21ES033118 (NIH)
Record Dates: First submitted 2022-01-10; First posted 2022-02-04 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Asthma; Environmental Exposure; Home Environment Related Disease
Keywords: volatile organic compounds; particulate matter; home air quality; asthma control; ecological momentary assessment; home air quality monitoring; smartphone technology; home spirometry
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Home Air Quality — This study will assess the feasibility and usability of ecological momentary assessment (EMA) to capture the context of real time behaviors and environmental exposures that impact indoor environments. In addition, the study will assess the feasibility and usability of providing participants with a readily available indoor home air quality monitor to continuously capture total volatile organic compounds (VOCs) and particulates (PM2.5).

SUMMARY:
The purposes of this study are to determine the practicality of using home indoor air quality monitoring and a smartphone app to identify home air quality changes and how these changes affect adults with asthma.

DETAILED DESCRIPTION:
The aims of this feasibility study are: 1) determine the feasibility and usability of: (a) ecological momentary assessment (EMA) to assess self-report residential environmental exposures and asthma symptoms, (b) home monitoring of objective environmental exposures (total volatile organic compounds [VOCs], particulates [PM2.5]), and lung function (home spirometry); 2a) assess the frequency and degree of residential environmental exposures (e.g., disinfectants/cleaners, second-hand smoke) via (a) self-reported data, and (b) home monitoring objective measures, 2b) assess the level of asthma control as indicated by self-reported asthma symptoms and lung function; and 3) explore associations of self-reported and objective measures of residential environmental exposures with self-reported and objective measures of asthma control. Participants will receive an indoor air quality monitor and a home spirometer to measure VOCs, PM2.5, and forced expiratory volume percent predicted, respectively. EMA will be collected using a personal smartphone and EMA software platform. Participants' will be sent scheduled and random EMA notifications to assess asthma symptoms, environmental exposures, lung function, and mitigation strategies. After the 14-day data collection period, participants will respond to survey items related acceptability, appropriateness, and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Adults who previously participated in the online Global Covid-19 and Asthma Study, indicated willingness to be contacted for future research, and reported high use of disinfectant/cleaning products since COVID-19 (≥5 per week).
* Current Asthma Control Test (ACT) ≤19
* Own a smartphone
* Have a Wi-Fi/wireless internet connection in their home.

Exclusion Criteria:

* Non-US residents
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with asthma living in the US
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Polivka, PhD, Principal Investigator — Select
Locations (1):
- Barbara J Polivka, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
To maximize the utility of this research, and in the interests of allowing other researchers and the public to benefit from it, the investigators will make the entire protocol and deidentified dataset available to researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Up to 24 months after the publication of the main study findings.
Access Criteria: Requests for IPD will be reviewed by the MPIs once a formal email request is submitted for research addressable aims/questions/hypotheses. Once the request has been approved by the MPIs and IRB approval is obtained, only deidentified data relevant to the research questions will be shared for secondary analyses deemed appropriate by the MPIs.
URL: https://www.kumc.edu/school-of-nursing/research.html

REFERENCES:
- [Background] Eldeirawi K, Huntington-Moskos L, Nyenhuis SM, Polivka B. Increased disinfectant use among adults with asthma in the era of COVID-19. J Allergy Clin Immunol Pract. 2021 Mar;9(3):1378-1380.e2. doi: 10.1016/j.jaip.2020.12.038. Epub 2020 Dec 29. No abstract available. PMID 33385592
- [Background] Matulonga B, Rava M, Siroux V, Bernard A, Dumas O, Pin I, Zock JP, Nadif R, Leynaert B, Le Moual N. Women using bleach for home cleaning are at increased risk of non-allergic asthma. Respir Med. 2016 Aug;117:264-71. doi: 10.1016/j.rmed.2016.06.019. Epub 2016 Jun 25. PMID 27492540
- [Background] Le Moual N, Varraso R, Siroux V, Dumas O, Nadif R, Pin I, Zock JP, Kauffmann F; Epidemiological Study on the Genetics and Environment of Asthma. Domestic use of cleaning sprays and asthma activity in females. Eur Respir J. 2012 Dec;40(6):1381-9. doi: 10.1183/09031936.00197611. Epub 2012 Apr 10. PMID 22496323
- [Background] Zock JP, Plana E, Jarvis D, Anto JM, Kromhout H, Kennedy SM, Kunzli N, Villani S, Olivieri M, Toren K, Radon K, Sunyer J, Dahlman-Hoglund A, Norback D, Kogevinas M. The use of household cleaning sprays and adult asthma: an international longitudinal study. Am J Respir Crit Care Med. 2007 Oct 15;176(8):735-41. doi: 10.1164/rccm.200612-1793OC. Epub 2007 Jun 21. PMID 17585104
- [Background] Gharpure R, Hunter CM, Schnall AH, Barrett CE, Kirby AE, Kunz J, Berling K, Mercante JW, Murphy JL, Garcia-Williams AG. Knowledge and Practices Regarding Safe Household Cleaning and Disinfection for COVID-19 Prevention - United States, May 2020. MMWR Morb Mortal Wkly Rep. 2020 Jun 12;69(23):705-709. doi: 10.15585/mmwr.mm6923e2. PMID 32525852
- [Derived] Nyenhuis S, Cramer E, Grande M, Huntington-Moskos L, Krueger K, Bimbi O, Polivka B, Eldeirawi K. Utilizing Real-time Technology to Assess the Impact of Home Environmental Exposures on Asthma Symptoms: Protocol for an Observational Pilot Study. JMIR Res Protoc. 2022 Aug 2;11(8):e39887. doi: 10.2196/39887. PMID 35916686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5/2022 to 2/2023. Eligibility criteria included previous participation in the Global COVID-19 and Asthma Study (GCAS), willingness to be contacted for future research, high use of disinfectant/cleaning products during COVID-19 (≥5 per week), Asthma Control Test score ≤19 or ≥2 asthma exacerbations in the previous 12 months, owned a smartphone, and had Wi-Fi/wireless connection in their home. Non-US residents and non-English speakers were excluded.
Groups:
- A Feasibility Study to Capture Residential Environmental Exposures and Asthma Symptoms in Adults: We assessed the feasibility and usability of ecological momentary assessment (EMA) to capture the context of real time behaviors and environmental exposures that impact indoor environments. In addition, we assessed the feasibility and usability of providing participants with a readily available indoor air quality monitor (Awair Omni®) to continuously capture total volatile organic compounds (VOCs) and particulates (PM2.5). This design will allowed us to alert participants of high levels and collect real time data on exposures and asthma symptoms. Daily and exposure-related lung function were measured with a low-cost home spirometer. Finally, we examined the effect of residential environmental exposures that may be related to increased time spent at home due to COVID-19 and the associations between these exposures and asthma control.
Period: Overall Study
Arm/Group | A Feasibility Study to Capture Residential Environmental Exposures and Asthma Symptoms in Adults
Started | 64
Completed | 40
Not Completed | 24
Not completed — Lost to Follow-up | 24

BASELINE CHARACTERISTICS:
Arm/Group | A Feasibility Study to Capture Residential Environmental Exposures and Asthma Symptoms in Adults
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 44
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Episodes Per Day
Description: Number of episodes per day that the residential VOCs exceeded 333 ppb and/or PM2.5 exceeded 15 mg/m3, as measured by the Awair home air quality monitor
Time Frame: Measured daily for 14 days
Measure: Mean (Standard Deviation); unit: Episodes per day
Arm/Group | A Feasibility Study to Capture Residential Environmental Exposures and Asthma Symptoms in Adults
Number analyzed (Participants) | 40
Episodes per day | 2.22 (1.41)

2. Primary Outcome: Home Spirometry Completed
Description: Number of participants completing daily home spirometry over 14 days.
Time Frame: Assessed daily for 14 days
Measure: Number; unit: participants
Groups:
- Arm 1: All participants completing feasibility study
Arm/Group | Arm 1
Number analyzed (Participants) | 40
participants | 40

3. Secondary Outcome: Integration of Study Components
Description: Participants were asked one survey item to assess if the various components of the study were well integrated. Response options ranged from 0=Strongly disagree to 4=Strongly agree. The score was multiplied by 25; scores could range from 0-100. A higher score indicated that the study components were well integrated.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1
Number analyzed (Participants) | 40
score on a scale | 87.2 (20.9)

4. Secondary Outcome: Ecological Momentary Assessment (EMA) Surveys
Description: Number of participants completing air quality triggered EMA surveys
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | A Feasibility Study to Capture Residential Environmental Exposures and Asthma Symptoms in Adults
Number analyzed (Participants) | 40
Participants | 40

ADVERSE EVENTS:
Time Frame: 14 days per participant
Arm/Group | A Feasibility Study to Capture Residential Environmental Exposures and Asthma Symptoms in Adults
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

LIMITATIONS AND CAVEATS:
This was a feasibility study with a small sample thus potentially limiting generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT05224076/Prot_SAP_000.pdf